CLINICAL TRIAL: NCT07188870
Title: Investigating the Prevalence and Associations of Autistic Traits, Feeding Difficulties, and Atypical Sensorimotor Integration in the Hungarian Early Childhood Population.
Brief Title: Associations of Autistic Traits and Feeding Difficulties
Acronym: BAMBI2025
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Gábor Csukly, Associate Professor, Semmelweis University
Other Study IDs: BAMBI2025
Record Dates: First submitted 2025-07-25; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BAMBI_pos: children with BAMBI scores higher than the cut-off
- BAMBI_neg: children with BAMBI scores lower than the cut-off

SUMMARY:
The objective is to assess the prevalence of autistic traits and feeding disorders in the general population.

DETAILED DESCRIPTION:
The objective of our research is twofold:

I. Firstly, the objective is to assess the prevalence of autistic traits and feeding disorders in the general population. The long-term goal is to develop a widely applicable screening tool for early autism detection that can be widely applied by primary care professionals.

1. To implement this survey, it is necessary to translate, adapt, and validate the screening instruments (questionnaires) into Hungarian.
2. The objective of the study is to administer the finalised version of the questionnaire to a large sample of parents, with a view to investigating the associations between autism and eating difficulties.

II. Secondly, in the clinical phase of our study, we aim to investigate in greater depth the relationship between feeding difficulties and autism spectrum disorder. In this phase, participants (children in the study group and their parents) will undergo in-person assessments and complete additional questionnaires:

1. For the objective observation of eating difficulties and autistic symptoms, as well as to compare these findings with earlier responses to the screening questionnaire;
2. To identify potential additional influencing factors, we will assess the child's somatic status and sensory sensitivities, as well as parental attitudes (e.g., anxiety, attachment, attitudes).

ELIGIBILITY:
Inclusion Criteria:

* Age between 1.5 and 6 years
* Diagnostic status:
* Diagnosed with autism spectrum disorder;
* Showing signs of ASD without formal diagnosis;
* Neurotypical development
* Children and their parents
* Parental consent to participate in the study

Exclusion Criteria:

* Developmental disorders affecting feeding
* Children living in institutional care separated from parents
* Medication affecting feeding behavior
* Malnutrition due to poverty
* Parents with low educational attainment or severe communication difficulties preventing questionnaire completion

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Questionnaires will be made available to parents of Hungarian children between 18 - 72 months, diagnosed with ASD by clinicians involved in their care. Parents of neurotypical or undiagnosed children will be reached through social media platforms and via family pediatricians and health visitors in primary care.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Brief Autism Mealtime Behavior Inventory "BAMBI"scores | Cross-sectional study. Through study completion, an average of two years.

CONTACTS AND LOCATIONS:
Locations (1):
- Bethesda Children's Hospital, Budapest, Hungary